CLINICAL TRIAL: NCT00006382
Title: Lung Screening Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000068258; NCI-LUNG; NCI-P00-0171
Record Dates: First submitted 2000-10-04; First posted 2004-06-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — X-Rays

INTERVENTIONS:
Procedure: bronchoscopic and lung imaging studies
Procedure: comparison of screening methods
Procedure: computed tomography
Procedure: radiography
Procedure: study of high risk factors

SUMMARY:
RATIONALE: New imaging procedures such as spiral CT may improve the ability to detect lung cancer in patients who are at high risk for the disease.

PURPOSE: Randomized clinical trial to compare the effectiveness of a spiral CT scan with that of a chest x-ray in detecting lung cancer in patients who are at high risk for the disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of screening spiral CT scan and screening chest x-ray in detecting lung cancer in current or former smokers at high risk for lung cancer.

OUTLINE: This is a randomized, multicenter study of lung cancer screening. Patients are randomized to one of two screening arms. Arm I: Patients undergo one spiral CT scan. Arm II: Patients undergo one chest x-ray. Patients and their primary care physicians are notified of test results within 3 weeks of the exam.

PROJECTED ACCRUAL: A total of 3,000 participants (1,500 per screening arm) will be accrued for this study at six screening centers (500 per center) by October 31, 2000.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: Age: 55 to 74 Patients with a cigarette smoking history of at least 30 pack-years Current smoker OR Smoker who has quit smoking within the past 10 years No known prior history of lung cancer

PRIOR CONCURRENT THERAPY: No concurrent therapy for any cancer except nonmelanomatous skin cancer No prior removal of any portion of the lungs No concurrent participation in other cancer screening trial, including PLCO No concurrent participation in a primary cancer prevention trial other than a smoking cessation trial

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K. Gohagan, PhD, FACE, Study Chair — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Marshfield Clinic, Marshfield, Wisconsin

REFERENCES:
- [Result] Croswell JM, Baker SG, Marcus PM, Clapp JD, Kramer BS. Cumulative incidence of false-positive test results in lung cancer screening: a randomized trial. Ann Intern Med. 2010 Apr 20;152(8):505-12, W176-80. doi: 10.7326/0003-4819-152-8-201004200-00007. PMID 20404381
- [Result] Gohagan J, Marcus P, Fagerstrom R, Pinsky P, Kramer B, Prorok P; Writing Committee, Lung Screening Study Research Group. Baseline findings of a randomized feasibility trial of lung cancer screening with spiral CT scan vs chest radiograph: the Lung Screening Study of the National Cancer Institute. Chest. 2004 Jul;126(1):114-21. doi: 10.1378/chest.126.1.114. PMID 15249451